CLINICAL TRIAL: NCT05047692
Title: A Dose Escalation, Multicenter, Open, Phase I Study to Assess the Safety and Immunogenicity of AdCLD-CoV19-1, a COVID-19 Preventive Vaccine in Healthy Volunteers.
Brief Title: Safety and Immunogenicity Study of AdCLD-CoV19-1: A COVID-19 Preventive Vaccine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellid Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: AdCLD-CoV19-1-001
Record Dates: First submitted 2021-09-14; First posted 2021-09-17 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Covid19
Keywords: COVID-19; Prevention; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — AdCLD-CoV19-1 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Low dose (Experimental): The subject will receive a single dose of AdCLD-CoV19-1(5.0x10^10VP) as an intramuscular injection.
  Interventions: Biological: AdCLD-CoV19-1
- Group 2: High dose (Experimental): The subject will receive a single dose of AdCLD-CoV19-1(1.0x10^11VP) as an intramuscular injection.
  Interventions: Biological: AdCLD-CoV19-1

INTERVENTIONS:
Biological: AdCLD-CoV19-1 — Replication deficient adenoviral vector based COVID-19 prevention vaccine containing recombinant gene of SARS-CoV-2 spike protein

SUMMARY:
This is a Phase 1 clinical trial to assess the safety and immunogenicity of AdCLD-CoV19-1 in healthy adults.

DETAILED DESCRIPTION:
This is a dose-escalation, multi-center, open-label, Phase 1 clinical trial. We assess the safety of AdCLD-CoV19-1 and immune responses against SARS-CoV-2. DSMB will evaluate safety when events occurred during the whole study period.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to agree informed consent and aged 19 to 64 years.
* The BMI index is 18.5 kg/m2 to 30.0 kg/m2.
* Able and willing to medically effective contraception during the whole study period.
* Agreement to refrain from blood donation during the whole study period.

Exclusion Criteria:

* Anyone deemed infected by COVID-19.
* Determined to be a close-contact of SARS-CoV-2 confirmed case or classified to symptomatic patient of COVID-19 prior to vaccination.
* Clinically significant abnormal ranges of laboratory measurement, ECG, Chest X-ray at screening visit.
* Positive in HIV, HBV, HCV test at screening visit.
* Acute fever(≥ 38℃) or suspected infectious disease, symptoms of infectious disease(cough, difficulty breathing, chills, muscle aches, headache, sore throat, loss of smell, or loss of taste, etc.) within 3 days prior to vaccination.
* Chronic respiratory disease: Asthma, chronic obstructive pulmonary disease, active tuberculosis, latent tuberculosis under treatment.
* Clinically significant active or any history of disease: Hepatobiliary system, kidney, central or peripheral nervous system (epilepsy, seizure, etc.), endocrine system (uncontrolled diabetes, hyperlipidemia, etc.), cardiovascular system (congestive heart failure, coronary artery disease, myocardial infarction, control Hypertension, etc.), blood tumor, urinary system, mental, musculoskeletal system, immune system (rheumatoid arthritis, systemic lupus erythematosus).
* Immunosuppressive disease including immunodeficiency disease.
* Scheduled to undergo any surgery during the whole study period.
* Healthcare worker who provide medical care to SARS-CoV-2 cases or occupationally in high risk for SARS-CoV-2 exposure during the whole study period.
* Prisoners or subjects who are compulsorily detained. (involuntary incarceration)
* History of SARS or MERS.
* Allergic reaction or hypersensitivity to any ingredient of AdCLD-CoV19-1.
* Having hemophilia at risk of causing serious bleeding when injected intramuscularly or receiving anticoagulants.
* Any history of malignant disease within the past 5 years. History of hypersensitivity to inoculate vaccine such as Guillain-Barre syndrome.
* History of serious adverse reaction or allergic reaction to inoculate vaccine.
* Urticaria past 5 years prior to vaccination.
* History of hereditary angioneurotic edema or acquired angioneurotic edema.
* History of solid organ or bone marrow transplantation.
* Suspected or a history of drug or alcohol abuse past 12 month before vaccination.
* Receipt of vaccine of SARS-CoV, MERS-CoV, SARS-CoV-2.
* Receipt of adenovirus vector based vaccine.
* Chronic use of immunosuppressant or immune modifying drug within 6 months prior to vaccination. (use of inhaled, topical, nasal, and ophthalmic corticosteroids are allowed)
* Having relied on antipsychotic drugs and narcotic analgesics within 6 months before vaccination or difficult to comply with the clinical trial procedure at the judgment of the investigator.
* Administered to other investigational product or medical device within 6 months before vaccination.
* Other vaccination history within 30 days prior to vaccination or being scheduled within 30 days after vaccination.
* Receipt of immunoglobulin or any blood product within 3 month prior to vaccination.
* Pregnant(including positive hCG test at screening visit) or breastfeeding female.
* Those who are directly related to the investigator.
* Other condition deemed ineligible for the study at the discretion of investigator.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited adverse events(AEs) | Through 7 days post-vaccination
Incidence of unsolicited AEs | Through 28 days post-vaccination

SECONDARY OUTCOMES:
Incidence of serious adverse events(SAEs) | Through 12 months post-vaccination
Incidence of adverse events of special interest(AESIs) | Through 12 months post-vaccination
Seroconversion rate(SCR) of neutralization antibody against wild type SARS-CoV-2 | 4 weeks post-vaccination
Geometric mean titer(GMT) of neutralization antibody against wild type SARS-CoV-2 | 4 weeks post-vaccination
GMT of S protein specific antibody | 2, 4, 26, 52 weeks post-vaccination
S protein specific T cell response | 2, 4, 26, 52 weeks post-vaccination

OTHER OUTCOMES:
GMT of S protein receptor binding domain(RBD) specific antibody | 2, 4, 26, 52 weeks post-vaccination

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Korea University Ansan Hospital, Ansan, Province
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon, Province
  - Korea University Guro Hospital, Seoul, State